CLINICAL TRIAL: NCT03015714
Title: Effectiveness of Aquatic Therapy for Parkinson's Disease Patients in the Context of a Multidisciplinary, Intensive Rehabilitation Treatment
Brief Title: Aquatic Therapy for Freezing of Gait in Parkinson's Disease Patients
Acronym: AT-FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: "Moriggia-Pelascini" Hospital
Record Dates: First submitted 2017-01-07; First posted 2017-01-10 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic; Gait Disorder, Sensorimotor
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIRT (Active Comparator): Patients in this group will undergo a 4-week Multidisciplinary Intensive Rehabilitation Treatment (MIRT).
  Interventions: Other: MIRT
- MIRT-AT (Active Comparator): Patients in this group will undergo a 4-week Multidisciplinary Intensive Rehabilitation Treatment associated with Aquatic Therapy (MIRT-AT).
  Interventions: Other: MIRT-AT

INTERVENTIONS:
Other: MIRT — MIRT consists of a 4-week rehabilitation program in a hospital setting, which entails four daily sessions of physical therapy for five days and one hour of physical exercise on the sixth day. On the seventh day the patient rests. The duration of each session, including recovery periods, is about one hour. The first session consists of a one-to-one session with a physical therapist. The second session includes aerobic exercises to improve balance and gait, using different devices: a stabilometric platform with visual cues, a treadmill plus and a cycloergometer. The third session consists of occupational therapy, the fourth one includes one hour of speech therapy.
  Arms: MIRT
Other: MIRT-AT — Patients in the MIRT-AT group will undergo the land-based therapy described in MIRT plus three sessions per week (Monday, Wednesday, Friday) of aquatic therapy. On days of aquatic therapy the first session of MIRT was not provided. The aquatic therapy program included aerobic exercises and physical activities to improve balance, motor skills, coordination and joints mobility. The water sessions were divided into 3 phases: i) Warm Up Exercises, ii) Central session Training, iii) Cool-down.
  Arms: MIRT-AT

SUMMARY:
Evaluation of the effectiveness of aquatic therapy for the treatment of freezing of gait in Parkinson's disease patients undergoing a multidisciplinary and intensive rehabilitation treatment.

DETAILED DESCRIPTION:
Freezing of gait (FoG) is an often dramatic, disabling episodic gait pattern that is common in Parkinson's disease (PD). FoG highly impairs mobility, causes falls, and reduces quality of life. Given the limited effectiveness of both the dopaminergic therapy and the deep brain stimulation on this symptom, it represents a challenge in the field of rehabilitation. In the last years, some studies described the effectiveness of aquatic therapy on balance dysfunction in patients with PD, correlating it to the safe conditions offered by the aquatic environment and to the physical properties of water. Nevertheless, the issues concerning the feasibility and the effectiveness of aquatic therapy for the treatment of FoG have never been addressed before. The aquatic environment may act on the sensorial peripheral receptors, thus widely stimulating the proprioceptive system. PD patients show an altered processing of the proprioceptive information that could potentially underline FoG. The investigators aim at investigating the effects of aquatic therapy for the treatment of FoG in PD patients undergoing a Multidisciplinary Intensive Rehabilitation Treatment (MIRT), whose effectiveness on several motor and functional parameters has been already demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to Gelb et al;
* Hoehn & Yahr (H&Y) stage 2.5-3;
* Presence of FOG confirmed in the patient assessment prior to participation in the study;
* Stable pharmacological treatment for the last 8 weeks and during the rehabilitation period;
* Mini Mental State Examination (MMSE) ≥ 24;

Exclusion Criteria:

* Cardiac, pulmonary, vestibular and orthopedic diseases;
* Urinary incontinence;
* Severe dyskinesias;
* Patients treated with deep brain stimulation;
* Visual deficits;
* Comorbilities other than PD determining reduction of motor autonomy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Freezing of Gait Questionnaire (FOGQ) | 4 weeks
  Assess FoG frequency, disturbances in gait and relationship to clinical features conceptually associated with gait and motor aspects.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale tot (UPDRS tot) | 4 weeks
  Clinician-scored monitored patient's global evaluation.
Unified Parkinson's Disease Rating Scale Part III (UPDRS III) | 4 weeks
  UPDRS subpart: clinician-scored monitored patient's motor evaluation
Unified Parkinson's Disease Rating Scale Part II (UPDRS II) | 4 weeks
  UPDRS subart: clinician-scored monitored patient's activitied daily life evaluation
Berg Balance Scale (BBS) | 4 weeks
  Motor-functional test for balance evaluation
Timed Up and Go Test (TUG) | 4 weeks
  Motor-functional test for sit to stand, walking and turning evaluation
Six Minutes Walking Test (6MWT) | 4 weeks
  Motor-functional test for gait endurance

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Study Director — "Moriggia-Pelascini" Hospital
Locations (1):
- "Moriggia-Pelascini" Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clerici I, Maestri R, Bonetti F, Ortelli P, Volpe D, Ferrazzoli D, Frazzitta G. Land Plus Aquatic Therapy Versus Land-Based Rehabilitation Alone for the Treatment of Freezing of Gait in Parkinson Disease: A Randomized Controlled Trial. Phys Ther. 2019 May 1;99(5):591-600. doi: 10.1093/ptj/pzz003. PMID 30657995